CLINICAL TRIAL: NCT02697890
Title: Effect of Mucograft® Seal on Post-extraction Ridge Preservation Using Bone Allograft: A Randomized Controlled Clinical Trial and Radiographic Evaluation
Brief Title: Effect of Mucograft® Seal on Post-extraction Ridge Preservation Using Bone Allograft
Acronym: Mucograft
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tufts University (Other)
Responsible Party: Principal Investigator, Natalie Jeong, Associate Professor, Tufts University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 11360
Record Dates: First submitted 2016-02-17; First posted 2016-03-03 (Estimated); Results first posted 2017-05-16 (Actual); Last update posted 2020-03-31 (Actual); Status verified 2020-03

CONDITIONS: Tooth Extraction Status Nos

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- FDBA (MinerOss®) + Collagen Sponge (HeliPLUG®) (Active Comparator): Interventions:
  Procedure: Ridge preservation procedure
  Interventions: Device: FDBA (MinerOss®) + Collagen Sponge (HeliPLUG®)
- FDBA (MinerOss®) + Mucograft® seal (Experimental): Interventions:
  Device: Mucograft® seal Procedure: Ridge preservation procedure
  Interventions: Device: FDBA (MinerOss®) + Mucograft® seal

INTERVENTIONS:
Device: FDBA (MinerOss®) + Mucograft® seal — Collagen matrix membrane for soft-tissue regeneration
  Arms: FDBA (MinerOss®) + Mucograft® seal
Device: FDBA (MinerOss®) + Collagen Sponge (HeliPLUG®) — Standard of Care
  Arms: FDBA (MinerOss®) + Collagen Sponge (HeliPLUG®)

SUMMARY:
The objective of this study is to evaluate clinically and radiographically the effect of Mucograft® seal when used for the ridge preservation procedure in combination with Freeze Dried Bone Allograft (FDBA) at the extraction site in terms of hard and soft tissue remodeling after 4 months healing period.

DETAILED DESCRIPTION:
One of the serious consequences of single or multiple tooth extraction is the bone resorption that follows, which may create aesthetic problems and compromise future implant placement. Ridge preservation procedures typically use a combination of a scaffold and a membrane. Scaffolds most commonly used are bone grafts; autogenous, allografts, xenografts, and alloplasts. Among these bone grafts, allograft materials such as Demineralized Freeze Dried Bone Allograft (DFDBA) and Freeze Dried Bone Allograft (FDBA) are frequently used in site preservation procedures.

An additional alternative is to use a collagen sponge (CS) in the extraction socket to prevent the infiltration of soft tissues to the lower area and to protect and maintain bone graft materials.

Although ridge preservation has several benefits, it also has several risks and limitations, such as membrane exposure and possible infection, loss or fibrous encapsulation of graft particles, longer healing period prior to implant placement, invasive and technique sensitive procedure, additional cost, and possible soft tissue dehiscence in bone grafted sites compared with non-grafted sites. Therefore, any modifications of the technique that will reduce these risks and limitations would be advantageous.

Mucograft® TM has been specifically designed for soft-tissue regeneration. Its bi-layer structure supports tissue in-growth and regeneration and promotes cellular and extracellular integration within the host tissue. Clinically, this new collagen membrane was associated with a sufficient width of newly formed attached gingiva with coverage of Miller class-I and class-II recession defects. These results suggest that the use of Mucograft® TM in periodontal plastic surgery may provide a viable source of grafting material as an alternative to autogenous and non-autogenous soft tissue graft materials.

This study is a clinical and radiographic, randomized parallel arm comparative evaluation of the addition of Mucograft® seal to FDBA in the ridge preservation procedure. Group A will receive FDBA and a CS. Group B will receive FDBA with Mucograft® seal.

ELIGIBILITY:
Inclusion Criteria:

* Be at least 18 years of age.
* Have unsalvageable non-adjacent non-molar teeth scheduled for extraction: maxillary incisors, canines, and premolars, and mandibular canines and premolars that require an extraction with ridge preservation planned for delayed implant placement. If a subject has multiple teeth to be extracted, only one tooth will be included in the study.
* Presence of buccal plate at the extraction site as determined by first sectional CBCT scan.
* Patients who are currently treatment planned in the Tufts University School of Dental Medicine (TUSDM) periodontology clinic to receive ridge preservation and meet all medical and dental requirements of the TUSDM periodontology clinic for periodontal surgery (e.g., subjects with no diseases or medication allergies contraindicating periodontal surgery).
* Display no evidence of acute periodontal infection: e.g., abscess, suppuration, severe swelling and/or spontaneous bleeding.
* Non-smoker or smoke less than 10 cigarettes per day.
* Not participating in any other research study for the duration of this study.

Exclusion Criteria:

* Have any known disease that interferes with periodontal surgery and would not allow the patient to be treatment planned for the procedures in the TUSDM periodontology clinic (e.g., severe anemia, low white blood cell count, bleeding or coagulation disorder, uncontrolled hypertension (150/90), recent myocardial infarction (within 6 months of enrollment), diabetes (HbA1C ≥7%), HIV/AIDS (self-reported), history of or currently undergoing head and neck radiation, history of or currently taking bisphosphonates, endocrine-induced bone diseases (e.g. hyperparathyroidism), immunosuppressive therapy).
* Have limited mental capacity and unable to give informed consent.
* Be a pregnant or lactating female (self-reported) (following TUSDM periodontology clinic guidelines elective surgical procedures and radiographs/CBCT scans are usually postponed until after delivery).
* Any known allergy/hypersensitivity to FDBA (contains trace amount of gentamicin, providone-iodine), CS or Mucograft® seal.
* Any known allergy to yeast.
* Have untreated acute infection at surgical site.
* Have untreated malignant neoplasm.
* Individuals opposed to having porcine derived materials placed in their mouth due to any personal reasons such as religious reasons.
* Teeth requiring flap reflection for extraction, e.g. deep subgingival caries or fractures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2015-05 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Natalie Jeong, DMD, Principal Investigator — Tufts University School of Dental Medicine

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- FDBA(MinerOss®) + Collagen Sponge(HeliPLUG®): Interventions:
  Procedure: Ridge preservation procedure
  FDBA (MinerOss®) + Collagen Sponge (HeliPLUG®): Standard of Care
- FDBA (MinerOss®) + Mucograft® Seal: Interventions:
  Device: Mucograft® seal Procedure: Ridge preservation procedure
  FDBA (MinerOss®) + Mucograft® seal: Collagen matrix membrane for soft-tissue regeneration
Period: Overall Study
Arm/Group | FDBA(MinerOss®) + Collagen Sponge(HeliPLUG®) | FDBA (MinerOss®) + Mucograft® Seal
Started | 14 | 14
Completed | 14 | 14
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | FDBA(MinerOss®) + Collagen Sponge(HeliPLUG®) | FDBA (MinerOss®) + Mucograft® Seal | Total
Number analyzed (Participants) | 14 | 14 | 28
Age, Continuous [Mean (Full Range); unit: years] | 55.6 [30 to 74] | 55.1 [25 to 80] | 55.4 [25 to 80]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 4 | 11
  Male | 7 | 10 | 17
Region of Enrollment [Number; unit: participants]
  United States | 14 | 14 | 28

OUTCOME MEASURES:

1. Primary Outcome: Changes in Alveolar Bone (mm)
Description: Width of Alveolar Bone at 4, 7, and 10mm heights apical to the CEJ buccally and lingually. Mean of overall buccal and lingual/palatal height (reference hole to buccal and lingual bone top).Assessed clinically by caliper/periodontal probe and radiographically by CBCT scans
Time Frame: 4 months after surgical procedure
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | FDBA(MinerOss®) + Collagen Sponge(HeliPLUG®) | FDBA (MinerOss®) + Mucograft® Seal
Number analyzed (Participants) | 14 | 14
mm | -1.47 (1.29) | -1.21 (1.22)

2. Secondary Outcome: Changes in Hard Tissues
Description: Clinical measurements will be recorded using the prefabricated stent and its horizontal and vertical reference holes along with a caliper.
Time Frame: 4 months after surgical procedure
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | FDBA(MinerOss®) + Collagen Sponge(HeliPLUG®) | FDBA (MinerOss®) + Mucograft® Seal
Number analyzed (Participants) | 14 | 14
mm | -0.79 (3.07) | -0.30 (1.09)

3. Secondary Outcome: Changes in Soft Tissues
Description: as for outcome 2
Time Frame: 4 months after surgical procedure
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | FDBA(MinerOss®) + Collagen Sponge(HeliPLUG®) | FDBA (MinerOss®) + Mucograft® Seal
Number analyzed (Participants) | 14 | 14
mm | 0.59 (1.28) | 0.90 (0.90)

4. Secondary Outcome: Keratinized Tissue Width (mm)
Description: Assessed clinically by caliper/periodontal probe and radiographically by CBCT scans.
Time Frame: 4 months after surgical procedure
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | FDBA(MinerOss®) + Collagen Sponge(HeliPLUG®) | FDBA (MinerOss®) + Mucograft® Seal
Number analyzed (Participants) | 14 | 14
mm | -0.08 (1.24) | -0.08 (0.54)

ADVERSE EVENTS:
Arm/Group | FDBA(MinerOss®) + Collagen Sponge(HeliPLUG®) | FDBA (MinerOss®) + Mucograft® Seal
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/14
Other Adverse Events (participants affected / at risk) | 0/14 | 0/14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No